CLINICAL TRIAL: NCT06838858
Title: Investigation of the Early Effects of Motor Imagery Training on Balance, Walking and Quality of Life After Ankle Plantar Flexor Muscle Lengthening Surgery in Children With Cerebral Palsy
Brief Title: Effects of Motor Imagery Training After Muscle Lengthening Surgery in Children With Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Meltem Çelik, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCDT-2025
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Rehabilitation; Cerebral Palsy (CP); Exercise; Tenotomy; Motor Imagery Training; Orthopedic Surgery
Keywords: Rehabilitation; Post-operative Rehabilitaton; Cerebral Palsy; Surgery; Tenotomy; Motor Imagery Training
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor Imagery Training Group in Addition to Post-Operative Exercise (Active Comparator): The study group will receive motor imagery exercises in addition to the post-op rehabilitation received by the comparison group. The exercises will given in a hibrit method (a face to face therapy session and 2 telerehabilitation session in an online platform in a week).
  The telerehabilitation sessions will given under the supervision of a remote physiotherapist. This group will take therapy sessions during 8 weeks. All the patients will have totally 8 face to face therapy sessions and 16 telerehabilitation sessions.
  Interventions: Procedure: Motor Imagery Training; Procedure: Conventional Post-operative Exercises
- Post-Operative Exercise Group (Active Comparator): This group will be included in a conventional post-operative rehabilitation program that includes intensive foot intrinsic muscle balance, bilateral ankle strengthening and range of motion exercises, and general body balance studies after plantar flexor muscle relaxation operations. In the rehabilitation program of the case group, exercises are planned under the supervision of a remote physiotherapist, with the telerehabilitation method (online live sessions) 2 days and 1 face to face therapy session will be done in a week. face therapy sessions and 16 telerehabilitation sessions.
  Interventions: Procedure: Conventional Post-operative Exercises

INTERVENTIONS:
Procedure: Motor Imagery Training — The study group will receive motor imagery training in addition to control group's exercise program. This process will proceed as follows; In motor imagery training videos taken with a 9-year-old healthy child will be watched.• The content of the videos will include exercises such as ankle dorsiflexion, heel tapping while walking, climbing and descending stairs, walking on a ramp, standing on a ramp, walking on soft ground, and walking on a treadmill.• The patients will watch these videos and then the relaxation, imagination and return to environment phases of motor imagery will be applied respectively.
  Arms: Motor Imagery Training Group in Addition to Post-Operative Exercise
Procedure: Conventional Post-operative Exercises — This group will receive conventional exercises in the post-op process. The exercises included in the conventional exercise program are;
  * Balance board exercises
  * Balance disc exercises
  * Bosu exercises
  * Balance pad exercises
  * Wobble board exercises
  * Walking on soft ground
  * Balance exercises on soft ground
  * Apraximations and tractions
  * Target angle exercise for ankle
  * General standing balance exercises (Eyes open and closed - single foot, double foot)
  * Ankle bidirectional ROM
  * Ankle bidirectional strengthening
  * Exercises to increase foot intrinsic muscle strength and balance
  * Functional exercises

SUMMARY:
In children with cerebral palsy (CP), spasticity occurs in the muscles due to upper motor neuron lesions. The muscle groups that are mostly spastic in the lower extremity are; the hip adductor and flexors, hamstrings, and ankle plantar flexors. Spasticity in the ankle plantar flexor muscles of these muscle groups causes contracture over time and restricts ankle dorsiflexion. Limitations in ankle dorsiflexion present as toe walking problems, balance loss, and various functional difficulties in children. Children with spasticity of the ankle plantar flexor muscles gastrocnemius and soleus are initially treated conservatively with exercise and positioning. However, after contracture occurs, treatment is performed using surgical methods. Surgical release of plantar flexor muscles is a method that has been proven to be effective and is frequently applied in the clinic. This surgery aims to remove the ankle dorsiflexion joint range of motion restriction, prevent toe walking, and improve the functional status of the child. However, since the plantar flexor muscles are in the antigravity muscle group, excessive release of these muscles can cause loss of balance and crouch gait. Therefore, it is important for this surgery to be performed by an experienced surgical team at the right time and to provide an exercise protocol aimed at stabilization by working both muscle groups in the postoperative period. In addition, after these surgeries, the patient is immobilized with a cast and orthosis for a while and the patient's active and passive movements are restricted with these devices. Motor Imagery; It is the process of learning a new movement or improving the quality of a known movement by visualizing it in a planned and intensive way in the mind of the person without performing any motor activity. This study hypothesized that the motor imagery training in the early rehabilitation process with movement restrictions after plantar flexor muscle relaxation operations will be effective on the patient's balance, walking, and quality of life.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a pathology that occurs as a result of a non-progressive lesion in the brain that develops due to various risk factors that may occur before, during, or after birth. The spastic type is the most common type of CP. Children with CP experience various problems in physical, psychological, mental, and social areas depending on the affected area of the brain and the degree of involvement. Motor function losses are the primary problem in individuals with CP. Children are classified according to the level of involvement with the gross motor function scale (GMFCS). While GMFCS level 1 indicates the mildest involvement, GMFCS level 5 indicates the most severe involvement.

Spasticity that occurs in the affected areas of the body after upper motor neuron lesions directly negatively affects the child's muscle and joint functions. The muscle groups where spasticity is commonly and frequently seen in the lower extremities are the hip adductor muscles, hamstrings, and ankle plantar flexor muscles. Ankle plantar flexor muscle spasticity can be seen in children of all GMFCS levels and negatively affects the child's functional status and reduces compliance with orthosis use. Increased ankle plantar flexor spasticity causes contracture in the ankle plantar flexors over time, which restricts ankle dorsiflexion. This condition often causes toe walking in children. Toe walking disrupts the child's general body balance and also negatively affects other upper segments, especially the knee joint.

The primary treatment option in the presence of ankle plantar flexor muscle spasticity is conservative treatment. Conservative treatment includes positioning the ankle in dorsiflexion and strengthening the dorsiflexor muscles, stretching the ankle plantar flexor muscles, performing relaxation exercises on the same muscle group, transferring weight in the appropriate position, and walking exercises.

In addition, in the presence of dynamic spasticity, the effectiveness of botulinum neurotoxin injection applied to the ankle plantar flexor muscles in cases where conservative treatment is inadequate has been shown in the literature. In cases where all these methods are inadequate, plantar flexor muscle contracture is present, and the child is functionally negatively affected, lengthening surgeries performed on the plantar flexor muscles are indicated. This operation can be performed only on the gastrocnemius muscle or on the Achilles tendon, which includes both the gastrocnemius and soleus muscles.

The ankle plantar flexor muscles are included in the antigravity muscle group and have an important role in general body balance. The length and strength of these muscles at a certain rate provide stabilization of the body segments. While the increased tone of these muscles disrupts this stabilization, the inability of the elongated muscle to provide sufficient core support after relaxations results in excessive dorsiflexion and suggests that it may cause walking problems and ultimately loss of balance. Therefore, when deciding on plantar flexor muscle relaxation operations applied to children with CP, it is thought that the right timing should be provided and the surgery should be performed with an experienced team in sufficient and correct amounts, and post-operative rehabilitation protocols that include intensive studies on gaining balance and stabilization in the post-operative period will increase balance and walking control.

Motor Imagery; It is the process of learning a new movement or increasing the quality of a known movement by visualizing it in a planned and intensive manner in the mind without performing any motor activity. In imagery, while not actually doing any activity; it is possible to experience it through mental imagery by seeing the image in the mind, feeling the movement as in the image, sensing the taste or smell of the image, and hearing its sound. The effectiveness of motor imagery training has been shown in children with CP. There is no study on its effectiveness in the postoperative period.

This study hypothesizes that motor imagery training, which will be applied in addition to the post-operative rehabilitation program, is effective on balance, walking, and quality of life, especially in children with CP, in the rehabilitation process where there is a mandatory restriction with plaster and orthosis after ankle plantar flexor muscle lengthening surgeries. The primary aim of this study is to examine the effect of motor imagery training, which will be applied in addition to post-operative rehabilitation after ankle plantar flexor muscle release operations in individuals with CP, on balance, gait, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with Cerebral Palsy
* Being between the ages of 7-18
* Being able to walk with or without support
* Not having received botulinum toxin injections into the ankle plantar flexor muscles in the last 6 months
* Being at the GMFCS level of 1,2 or 3
* Having an indication for ankle muscle release surgery and having a surgical plan
* Being receiving a developmental rehabilitation program
* Being able to follow given commands

Exclusion Criteria:

* Having dyskinetic, ataxic or hypotonic involvement
* Having any neurosurgery before
* Having any bone surgery for the foot or ankle before
* Having a bone surgery in the same session
* Mental retardation and not being able to take commands

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Range of Motion Measurement | Baseline, week 4, week 8
  Range of Motion will be measured with using an universal goniometer for knee and ankle.
Muscle Strength | Baseline, week 4, week 8
  Manuel muscle testing will be done. It will graded 0 to 5. Five represents full strength.
Gait Assessment | Baseline and week 8
  It will be asseessed with using Edinburg Visual Gait Scorring (EVGS). EVGS is a video based gait scorring system. It consist of 17 items. A gait video will be taken from sagital and coronal plan. It will scorred later.
  Additionally, pedobarographic measurements for temporospatial gait parameters will be obtained with Enertor foot scanning system (RSscan Lab Ltd; UK).
  The temporospatial gait parameters are; step length, stride length, Step width, cadance, double support time, single support time.
Balance Assessment | Baseline, week 8
  It will done by using Pediatric Balance Scale. There are 14 items in this scale. The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills during tasks that mimic experiences of everyday living in school-aged children. The scale consists of 14 balance-related test items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
  Additionally, pedobarographic measurements for static balance assessment will be obtained with Enertor foot scanning system (RSscan Lab Ltd; UK).
Quality of Life Assessment | Baseline and week 8
  Quality of life assessments of patients will be made using the Quality of Life Scale for Children. The first version of the scale (PedsQL TM 1.0) is a general quality of life scale developed for use in various pediatric populations. The most powerful version, the fourth version's core scale (PedsQL TM 4.0 Generic Core Scale), is a scale that evaluates the basic physical, mental and social health components determined by the World Health Organization in healthy children or those with acute or chronic diseases, together with school functionality. This scale consists of a total of 23 items and 4 subscales, including 8 items measuring physical functionality, 5 items measuring emotional functionality, 5 items measuring social functionality and 5 items evaluating school functionality.

SECONDARY OUTCOMES:
Functional Mobility | Baseline, week 4, week 8
  Functional status and ambulation assessment of patients will be made with the Functional Mobility Scale (FMS). The Functional Mobility Scale is a scale that evaluates how patients walk 5, 50 and 500 meters and ultimately divides them into 6 groups.
Foot pressure measurement | Baseline and week 8
  The pedobarograph is a device displaying and recording the instantaneous distribution of the pressure under the entire surface of the soles of the feet. The subject stands or walks on a transparent plate, in which light is conducted by total internal reflections. For the assessment of foot pressure, pedobarographic measurements will be obtained with the Enertor foot scanning system (RSscan Lab Ltd; UK).
Movement imagery | Baseline, week 8
  It will be assessed by usisng Movement imagery questionnaire for children-MIQ-C. This questionnaire was used to measure visual (internal, external skills) and kinesthetic imagery. It contains a total of 12 items, 4 items internal, 4 items external, and 4 items kinesthetic imagery skills. Within the scope of the questionnaire, the individual is asked to imagine 4 different movements from 3 different visual perspectives. During this test applied with the evaluator, the individual is asked to do the movement in the instructions once in reality and then to imagine doing the movement, and the clarity of this imagery is scored using a Likert-type scale between 1 (very difficult to feel) and 7 (very easy to feel). The questionnaire was developed by Martini et al..
Motor Imagery Training Fun and Clarity | After each therapy sessions
  An additional evaluation will be made with the Motor Imagery Training Fun and Clarity Scale. The fun level of motor imagery sessions and imagery training for individuals will be evaluated using a 0-10 point numerical rating scale (fun scale). There will be numbers from 0 to 10 on a 10 cm horizontal line. On the scale, 0 on the line means "not fun at all" and 10 means "very fun". The degree of fun will be recorded numerically between 0 and 10. Similarly, how clearly they can visualize the tasks imagined during the imagery sessions will be evaluated with a 0-10 point numerical rating scale (clarity scale). Individuals will be asked to evaluate clarity by stating that 0 on a 10 cm horizontal line means that imagery is not clear at all, and 10 means it is very clear.

CONTACTS AND LOCATIONS:
Overall Officials: Zuhal Didem Takinacı, PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartrick CT, Kovan JP, Shapiro S. The numeric rating scale for clinical pain measurement: a ratio measure? Pain Pract. 2003 Dec;3(4):310-6. doi: 10.1111/j.1530-7085.2003.03034.x. PMID 17166126
- [Background] 29. Crichton, N. (2001). Visual analogue scale (VAS). J Clin Nurs, 10(5), 706-6.
- [Background] 28. Doussoulin, A., & Rehbein, L. (2011). Motor imagery as a tool for motor skill training in children. Motricidade, 7(3), 37-43.
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Ottenbacher KJ, Taylor ET, Msall ME, Braun S, Lane SJ, Granger CV, Lyons N, Duffy LC. The stability and equivalence reliability of the functional independence measure for children (WeeFIM). Dev Med Child Neurol. 1996 Oct;38(10):907-16. doi: 10.1111/j.1469-8749.1996.tb15047.x. PMID 8870612
- [Background] Xu C, Wen XX, Huang LY, Shang L, Cheng XX, Yan YB, Lei W. Normal foot loading parameters and repeatability of the Footscan(R) platform system. J Foot Ankle Res. 2017 Jul 17;10:30. doi: 10.1186/s13047-017-0209-2. eCollection 2017. PMID 28725271
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Graham HK, Harvey A, Rodda J, Nattrass GR, Pirpiris M. The Functional Mobility Scale (FMS). J Pediatr Orthop. 2004 Sep-Oct;24(5):514-20. doi: 10.1097/00004694-200409000-00011. PMID 15308901
- [Background] 22. Abd El-Raheem, R. M., Kamel, R. M., & Ali, M. F. (2015). Reliability of using Kinovea program in measuring dominant wrist joint range of motion. Trends in Applied Sciences Research, 10(4), 224.
- [Background] Read HS, Hazlewood ME, Hillman SJ, Prescott RJ, Robb JE. Edinburgh visual gait score for use in cerebral palsy. J Pediatr Orthop. 2003 May-Jun;23(3):296-301. PMID 12724590
- [Background] Rodda JM, Graham HK, Carson L, Galea MP, Wolfe R. Sagittal gait patterns in spastic diplegia. J Bone Joint Surg Br. 2004 Mar;86(2):251-8. doi: 10.1302/0301-620x.86b2.13878. PMID 15046442
- [Background] 19. Palisano, R., Rosenbaum, P., Bartlett, D., Livingston, M., Walter, S., & Russell, D. (2007). GMFCS-E&R. CanChild Centre for Childhood Disability Research, McMaster University, 200(7).
- [Background] Verschuren O, Ketelaar M, Takken T, Van Brussel M, Helders PJ, Gorter JW. Reliability of hand-held dynamometry and functional strength tests for the lower extremity in children with Cerebral Palsy. Disabil Rehabil. 2008;30(18):1358-66. doi: 10.1080/09638280701639873. PMID 18850351
- [Background] Boone DC, Azen SP, Lin CM, Spence C, Baron C, Lee L. Reliability of goniometric measurements. Phys Ther. 1978 Nov;58(11):1355-60. doi: 10.1093/ptj/58.11.1355. PMID 704684
- [Background] 15. Cohen, J, (1988), Statistical Power Analysis for the behavioral sciences, 2. Edition, Taylor & Francis INC, New York, US.)
- [Background] Steenbergen B, Craje C, Nilsen DM, Gordon AM. Motor imagery training in hemiplegic cerebral palsy: a potentially useful therapeutic tool for rehabilitation. Dev Med Child Neurol. 2009 Sep;51(9):690-6. doi: 10.1111/j.1469-8749.2009.03371.x. PMID 19709140
- [Background] Decety J. The neurophysiological basis of motor imagery. Behav Brain Res. 1996 May;77(1-2):45-52. doi: 10.1016/0166-4328(95)00225-1. PMID 8762158
- [Background] Kay RM, Rethlefsen SA, Ryan JA, Wren TA. Outcome of gastrocnemius recession and tendo-achilles lengthening in ambulatory children with cerebral palsy. J Pediatr Orthop B. 2004 Mar;13(2):92-8. doi: 10.1097/00009957-200403000-00006. PMID 15076586
- [Background] Ruzbarsky JJ, Scher D, Dodwell E. Toe walking: causes, epidemiology, assessment, and treatment. Curr Opin Pediatr. 2016 Feb;28(1):40-6. doi: 10.1097/MOP.0000000000000302. PMID 26709689
- [Background] Cottalorda J, Gautheron V, Metton G, Charmet E, Chavrier Y. Toe-walking in children younger than six years with cerebral palsy. The contribution of serial corrective casts. J Bone Joint Surg Br. 2000 May;82(4):541-4. doi: 10.1302/0301-620x.82b4.10188. PMID 10855878
- [Background] Tardieu C, Lespargot A, Tabary C, Bret MD. Toe-walking in children with cerebral palsy: contributions of contracture and excessive contraction of triceps surae muscle. Phys Ther. 1989 Aug;69(8):656-62. doi: 10.1093/ptj/69.8.656. PMID 2748720
- [Background] Schlough K, Andre K, Owen M, Adelstein L, Hartford MC, Javier B, Kern R. Differentiating Between Idiopathic Toe Walking and Cerebral Palsy: A Systematic Review. Pediatr Phys Ther. 2020 Jan;32(1):2-10. doi: 10.1097/PEP.0000000000000659. PMID 31842091
- [Background] Yan Y, Fu X, Xie X, Ji S, Luo H, Yang F, Zhang X, Yang S, Xie P. Hip Adductor Intramuscular Nerve Distribution Pattern of Children: A Guide for BTX-A Treatment to Muscle Spasticity in Cerebral Palsy. Front Neurol. 2019 Jun 14;10:616. doi: 10.3389/fneur.2019.00616. eCollection 2019. PMID 31258508
- [Background] Bar-On L, Molenaers G, Aertbelien E, Van Campenhout A, Feys H, Nuttin B, Desloovere K. Spasticity and its contribution to hypertonia in cerebral palsy. Biomed Res Int. 2015;2015:317047. doi: 10.1155/2015/317047. Epub 2015 Jan 11. PMID 25649546
- [Background] Compagnone E, Maniglio J, Camposeo S, Vespino T, Losito L, De Rinaldis M, Gennaro L, Trabacca A. Functional classifications for cerebral palsy: correlations between the gross motor function classification system (GMFCS), the manual ability classification system (MACS) and the communication function classification system (CFCS). Res Dev Disabil. 2014 Nov;35(11):2651-7. doi: 10.1016/j.ridd.2014.07.005. Epub 2014 Jul 23. PMID 25062096
- [Background] Papavasiliou AS. Management of motor problems in cerebral palsy: a critical update for the clinician. Eur J Paediatr Neurol. 2009 Sep;13(5):387-96. doi: 10.1016/j.ejpn.2008.07.009. Epub 2008 Sep 7. PMID 18778959
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461